CLINICAL TRIAL: NCT06715930
Title: Nomogram for Predicting In-stent Stenosis After Pipeline Embolization Device Treatment in Patients with Intracranial Aneurysm: a Multicenter, Retrospective Model Development and Validation Study
Brief Title: Nomogram for Predicting In-stent Stenosis After Pipeline Embolization Device Treatment in Patients with Intracranial Aneurysm
Acronym: PED-ISS
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University International Hospital (Other)
Responsible Party: Principal Investigator, Ming Lv, MD, Beijing Tiantan Hospital
Other Study IDs: PED-ISS
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial aneurysm; In-stent stenosis; Pipeline embolization device; Nomogram
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ISS group: Patients presenting with in-stent stenosis (ISS) at imaging follow-up. ISS was defined as a growth process exceeding the limits of metal mesh, as evidenced by a visible gap between the contrast-filled vascular lumen and the internal contours of the pipeline embolization device.
  Interventions: Procedure: Interventional treatment
- Non-ISS group: Patients withou in-stent stenosis (ISS) at imaging follow-up. ISS was defined as a growth process exceeding the limits of metal mesh, as evidenced by a visible gap between the contrast-filled vascular lumen and the internal contours of the pipeline embolization device.
  Interventions: Procedure: Interventional treatment

INTERVENTIONS:
Procedure: Interventional treatment — The procedure was performed via the traditional transfemoral arterial approach, under general anesthesia and complete heparin anticoagulation. PEDs were introduced using Marksman or Phenom-27 microcatheters (Medtronic, Irvine, USA), while coils were introduced via Echelon-10 microcatheters (Medtronic, Dublin, Ireland). An appropriate working projection was used to generate three-dimensional rotational angiography. Un-subtracted images were used to verify whether PED was completely deployed and attached to the parent artery. Wall apposition was enhanced using balloon angioplasty if post-deployment imaging indicated inadequate apposition. Overlapping devices were used when a single PED was not enough to cover the aneurysm neck and reconstruct blood flow. Neurointerventionalists with more than 15 years of experience conducted all endovascular procedures. The same dual-antiplatelet therapy was used for 6 months post-procedure, followed by aspirin monotherapy for a minimum of 12 months.

SUMMARY:
Intracranial aneurysms (IAs) are the primary cause of non-traumatic subarachnoid hemorrhage with high morbidity and mortality. Flow diverters, such as pipeline embolization devices (PEDs), are among the most effective methods for treating IAs in recent years due to the maturity of interventional devices and minimally invasive techniques. Unlike conventional stents, PEDs modify the hemodynamics within the parent artery and aneurysm sac, allowing blood flow from the aneurysm sac, thus facilitating endothelialization of the aneurysm neck. As a result, aneurysms are completely removed from circulation with time. However, about 5.1%-38.5% of IA patients develop in-stent stenosis (ISS) even after successful PED implantation. ISS increases the risk of retreatment and ischemic complications, thereby affecting the long-term prognosis of IA patients. Therefore, preoperative determination of the patient's suitability for PED implantation can enhance patient-centered decision-making and improve the long-term prognosis of IA patients.

Although previous studies have evaluated the correlation between certain individual variables and ISS, there are few comprehensive models predicting ISS after PED treatment. Nomograms have been widely used for prediction of tumor survival and cardiovascular events. Nomograms incorporate multiple risk factors for predicting the patient's potential prognosis based on their individual risks. This study aimed to identify the predictors for ISS after PED treatment and to create and verify a nomogram for assessing individual risk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged18 to 75 years;
2. IAs patients treated with PEDs;
3. patients whose parent artery did not have significant atherosclerotic stenosis;
4. patients who had at least one digital subtraction angiography (DSA) follow-up.

Exclusion Criteria:

1. Patients missing critical clinical baseline;
2. patients with inadequate DSA image quality for reliable assessment;
3. patients with comorbid cerebrovascular conditions, including arteriovenous fistulas and arteriovenous malformations;
4. patients without any follow-up information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosis of "unruptured intracranial aneurysm" treated with PEDs.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
In-stent stenosis | 6 months, 1 year, and 3 years after treatment.
  In-stent stenosis was defined as a growth process exceeding the limits of metal mesh, as evidenced by a visible gap between the contrast-filled vascular lumen and the internal contours of the PED.

SECONDARY OUTCOMES:
Complete occlusion at the last angiographic follow-up | 6 months, 1 year, and 3 years after treatment
  At follow-up, the patient's aneurysm was completely occluded, with an OKM score of grade D.
  O'Kelly-Marotta grading scale was used to assess aneurysm occlusion status following PED treatment. Grade D indicated complete occlusion, while grades A, B, and C represented incomplete occlusion
Procedure-related complications | 6 months, 1 year, and 3 years after treatment
  Procedure-related complications were divided into hemorrhagic, ischemic, and compression symptoms. Hemorrhagic complications were defined as subarachnoid hemorrhage or distal intraparenchymal hemorrhage after PED implantation. Ischemic complications included in-stent thrombosis, transient ischemic attack, or cerebral infarction associated with the treated vascular area. Compression symptoms included neurological symptoms or brain stem symptoms associated with aneurysm compression.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turhon M, Kang H, Liu J, Zhang Y, Zhang Y, Huang J, Wang K, Li M, Liu J, Zhang H, Li T, Song D, Zhao Y, Luo B, Maimaiti A, Aisha M, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X, Guan S. In-Stent Stenosis After Pipeline Embolization Device in Intracranial Aneurysms: Incidence, Predictors, and Clinical Outcomes. Neurosurgery. 2022 Dec 1;91(6):943-951. doi: 10.1227/neu.0000000000002142. Epub 2022 Sep 21. PMID 36129281
- [Background] John S, Bain MD, Hui FK, Hussain MS, Masaryk TJ, Rasmussen PA, Toth G. Long-term Follow-up of In-stent Stenosis After Pipeline Flow Diversion Treatment of Intracranial Aneurysms. Neurosurgery. 2016 Jun;78(6):862-7. doi: 10.1227/NEU.0000000000001146. PMID 26600281
- [Background] Wang T, Richard SA, Jiao H, Li J, Lin S, Zhang C, Wang C, Xie X, You C. Institutional experience of in-stent stenosis after pipeline flow diverter implantation: A retrospective analysis of 6 isolated cases out of 118 patients. Medicine (Baltimore). 2021 Mar 19;100(11):e25149. doi: 10.1097/MD.0000000000025149. PMID 33725998
- [Background] Dong L, Wang C, Chen X, Li M, Li T, Liu H, Zhao Y, Duan R, Jin W, Zhang Y, Wang Y, Lv M. Predicting Persistent Aneurysm Filling After Pipeline Embolization Device Treatment in Patients with Intracranial Aneurysm: Development and External Validation of a Nomogram Model. Transl Stroke Res. 2025 Apr;16(2):392-402. doi: 10.1007/s12975-023-01222-9. Epub 2023 Dec 8. PMID 38066403
- [Background] Kadirvel R, Ding YH, Dai D, Rezek I, Lewis DA, Kallmes DF. Cellular mechanisms of aneurysm occlusion after treatment with a flow diverter. Radiology. 2014 Feb;270(2):394-9. doi: 10.1148/radiol.13130796. Epub 2013 Oct 28. PMID 24086073
- [Background] Kang H, Zhou Y, Luo B, Lv N, Zhang H, Li T, Song D, Zhao Y, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X, Liu J. Pipeline Embolization Device for Intracranial Aneurysms in a Large Chinese Cohort: Complication Risk Factor Analysis. Neurotherapeutics. 2021 Apr;18(2):1198-1206. doi: 10.1007/s13311-020-00990-8. Epub 2021 Jan 14. PMID 33447904
- [Background] Becske T, Kallmes DF, Saatci I, McDougall CG, Szikora I, Lanzino G, Moran CJ, Woo HH, Lopes DK, Berez AL, Cher DJ, Siddiqui AH, Levy EI, Albuquerque FC, Fiorella DJ, Berentei Z, Marosfoi M, Cekirge SH, Nelson PK. Pipeline for uncoilable or failed aneurysms: results from a multicenter clinical trial. Radiology. 2013 Jun;267(3):858-68. doi: 10.1148/radiol.13120099. Epub 2013 Feb 15. PMID 23418004
- [Background] Hanel RA, Cortez GM, Lopes DK, Nelson PK, Siddiqui AH, Jabbour P, Mendes Pereira V, Istvan IS, Zaidat OO, Bettegowda C, Colby GP, Mokin M, Schirmer CM, Hellinger FR, Given C, Krings T, Taussky P, Toth G, Fraser JF, Chen M, Priest R, Kan P, Fiorella D, Frei D, Aagaard-Kienitz B, Diaz O, Malek AM, Cawley CM, Puri AS, Kallmes DF. Prospective study on embolization of intracranial aneurysms with the pipeline device (PREMIER study): 3-year results with the application of a flow diverter specific occlusion classification. J Neurointerv Surg. 2023 Mar;15(3):248-254. doi: 10.1136/neurintsurg-2021-018501. Epub 2022 Mar 15. PMID 35292570
- [Background] Thompson BG, Brown RD Jr, Amin-Hanjani S, Broderick JP, Cockroft KM, Connolly ES Jr, Duckwiler GR, Harris CC, Howard VJ, Johnston SC, Meyers PM, Molyneux A, Ogilvy CS, Ringer AJ, Torner J; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention; American Heart Association; American Stroke Association. Guidelines for the Management of Patients With Unruptured Intracranial Aneurysms: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Aug;46(8):2368-400. doi: 10.1161/STR.0000000000000070. Epub 2015 Jun 18. PMID 26089327
- [Background] Liu Q, Li K, He H, Miao Z, Cui H, Wu J, Ding S, Wen Z, Chen J, Lu X, Li J, Zheng L, Wang S. The markers and risk stratification model of intracranial aneurysm instability in a large Chinese cohort. Sci Bull (Beijing). 2023 Jun 15;68(11):1162-1175. doi: 10.1016/j.scib.2023.05.001. Epub 2023 May 10. PMID 37210332